CLINICAL TRIAL: NCT03782844
Title: Efficacy of Simple Continuous Positive Airway Pressure on Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Key Laboratory of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Yuan-Ming Luo, Professor, State Key Laboratory of Respiratory Disease
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2011 No. 5
Record Dates: First submitted 2018-11-05; First posted 2018-12-20 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Sleep Apnea, Obstructive; Continuous Positive Airway Pressure; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional fixed CPAP and simple CPAP (Experimental): Participants in this group were manually titrated . They were treated with conventional fixed pressure CPAP and Simple CPAP for two separate nights in random order monitored by full polysomnography.
  Interventions: Device: Simple CPAP+Conventional fixed CPAP
- Auto CPAP and simple CPAP (Experimental): Participants in this group after being manually titrated were treated with Auto RemStar CPAP and Simple CPAP for two separate nights in random order monitored by full polysomnography.
  Interventions: Device: Simple CPAP + Auto CPAP

INTERVENTIONS:
Device: Simple CPAP+Conventional fixed CPAP — Patients used simple CPAP and conventional fixed CPAP during overnight polysomnography.
  Arms: Conventional fixed CPAP and simple CPAP
Device: Simple CPAP + Auto CPAP — Patients used simple CPAP and Auto CPAP during overnight polysomnography.
  Arms: Auto CPAP and simple CPAP

SUMMARY:
Obstructive sleep apnea (OSA) is a common and frequently-occurring disease. The incidence of OSA is more than 4% in general population, and as high as 20% - 40% in the elderly. At present, CPAP machines commonly used for OSA treatment includes traditional pressure fixed single-level CPAP machine and automatic pressure regulation CPAP machine. Studies have shown that the CPAP treatment pressure of OSA patients is normally below 11 cmH2O. Since the condition of OSA patients and the required CPAP treatment pressure may change over time, a CPAP machine with automatic pressure regulation function may theoretically better meet the needs of treatment. However, a recent large-scale clinical study with an average follow-up of four years showed that there was little need to change CPAP treatment pressure after titration. Although different types of CPAP have different functions, the basic principle is to keep the upper airway open and unobstructed to eliminate sleep apnea and hypopnea by continuously applying positive pressure to the upper respiratory tract through an air pump. A complex CPAP machine with functions such as pressure regulation, boost delay, end-expiratory pressure release will cost more than a single-function CPAP machine. Some patients from poor areas, even with severe OSA, may give up treatment when they can not afford CPAP machines that have not yet been included in national health insurance in China. In view of the current economic level in China, it is urgent to find an inexpensive and effective CPAP machine for the treatment of OSA and related complications. Recently, Guangzhou Yinghui Medical Technology Co., Ltd.and State Key Laboratory of Respiratory Disease have developed a new simple CPAP machine. The CPAP treatment pressure is fixed at the factory to 6 cm H2O (SKL), 8 cm H2O (SKM) and 10 cm H2O (SKH). Compared to traditional CPAP machine, only a power switch button is attached on the body, and the additional adjustment devices including display screen are removed, which not only reduces the cost of the CPAP machine, but also facilitates the operation of patients.

DETAILED DESCRIPTION:
Study Design: A randomized, cross-over and double blind study . Objective: To investigate the efficacy of simple device of continuous positive airway pressure (CPAP) in the treatment of obstructive sleep apnea (OSA). Methods: A randomized, cross-over and double blind study would be performed on 100 OSA patients using both simple CPAP and traditional CPAP during overnight polysomnography. Pressure for CPAP treatment would be manual titrated. The sleep apnea hypopnea index (AHI), arousal index (ArI), Oxygen desaturation Index (ODI), sleep structure and the preference of CPAP model were to be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate after informed consent
2. Males and females, any race and aged≥18yeras
3. Objectively confirmed OSA with an apnoea-hypopnoea- index (AHI)≥5/h by overnight polysomnography

Exclusion Criteria:

1. Central Sleep Apnoea/Cheyne Stokes Respiration
2. Opioid or sedative use; Alcohol abuse
3. Nasal congestion or tonsils more than Ⅱ degrees enlarged
4. Optimal treatment CPAP pressure over 10cmH2O
5. Poor understanding or being disabled

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | One full night
  Total number of apneas and hypopneas×60/total sleep time
Arousal Index | One full night
  Total number of arousals×60/total sleep time
Oxygen Desaturation Index | One full night
  Total number of oxygen desaturations≥3%×60/total sleep time
Sleep structure | One full night
  Sleep stage distribution(N1, N2, N3, NREM)
Adverse effects | Onefull night
  Using questionnaire to assess adverse effects including dyspnea, noise, bloating, et al

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided